CLINICAL TRIAL: NCT04577677
Title: Understanding the Neural Mechanisms Behind Transcranial Direct Current Stimulation
Brief Title: Understanding the Neural Mechanisms Behind tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Myles Mc Laughlin, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: S63709
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: tDCS Mechanisms
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- optimization of control anesthetic condition (Experimental)
  Interventions: Device: brain stimulation
- understanding tDCS effect on motor learning (Experimental)
  Interventions: Device: brain stimulation
- understanding tDCS effects on cortical excitability (Experimental)
  Interventions: Device: brain stimulation
- optimizing peripheral nerve stimulation protocols (Experimental)
  Interventions: Device: brain stimulation
- Effect peripheral nerve stimulation on motor learning (Experimental)
  Interventions: Device: brain stimulation

INTERVENTIONS:
Device: brain stimulation — tDCS and peripheral nerve stimulation
  Other Names: skin intervention

SUMMARY:
The aim of the study is to investigate the neural mechanisms underpinning transcranial direct current stimulation (tDCS), a non-invasive neuromodulation technique in which a direct current is passed through scalp electrodes. A series of experiments will be conducted to understand and characterize the transcranial and transcutaneous mechanisms of tDCS. To investigate this research question, every participant will undergo three stimulation conditions (active, sham and control). In the control condition, an anaesthetic cream will be applied to anaesthetize the nerves in the scalp. In addition, the effectiveness of tDCS and peripheral nerve stimulation will be compared. Ultimately, the obtained knowledge can lead to the development of improved non-invasive neuromodulation therapies, which can lead to more effective treatments of a variety of neurological and psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* good general health

Exclusion Criteria:

* Epilepsy or family history of epilepsy
* Migraine
* Allergic to lidocaine or benzocaine
* Pregnant
* History of or currently suffering from:
* neurological diseases
* psychiatric diseases, depression or anxiety (Annex B and Annex C)
* History of:
* brain surgery
* brain thrombosis
* cerebral hemorrhage
* severe head trauma
* meningitis
* long period of loss of consciousness (> 1 hour)
* Metal parts in the head or upper body:
* Defibrillator, implanted medication pump
* Metal prosthesis in ear, hart, …
* Deep brain stimulator
* Coronary bypass or intracranial or aneurysm clips (brain arteries, aorta, etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 30 minutes during stimulation
  Rate sensation from 0 ('I feel nothing') to 10 ('Stimulation is painful')
Reaction time | 20 minutes during tDCS stimulation
  Reaction time on the motor learning task
Reaction time | 20 minutes during peripheral nerve stimulation
  Reaction time on motor learning task
Amplitudes of event related potentials | during tDCS
  ERP during stimulation
Amplitudes of event related potentials | during peripheral nerve stimulation
  ERP during stimulation
Pupil dilations | during peripheral nerve stimulation
  pupil diameter during stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Seminck N, Van Bogaert T, Kilic U, Nuttin B, Mc Laughlin M. External Trigeminal Nerve Stimulation Evokes Bilateral Electroencephalography Responses and Modulates Spectral Power in Healthy Adults. Neuromodulation. 2025 Dec 26:S1094-7159(25)01146-8. doi: 10.1016/j.neurom.2025.11.002. Online ahead of print. PMID 41454900
- [Derived] Kerstens S, Orban de Xivry JJ, Mc Laughlin M. A novel tDCS control condition using optimized anesthetic gel to block peripheral nerve input. Front Neurol. 2022 Nov 14;13:1049409. doi: 10.3389/fneur.2022.1049409. eCollection 2022. PMID 36452171